CLINICAL TRIAL: NCT03121989
Title: Study to Evaluate the Feasibility of 13-C Pyruvate Imaging in Breast Cancer Patients Receiving Neoadjuvant Chemotherapy
Acronym: LABC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding completed
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 254-2015
Record Dates: First submitted 2017-02-10; First posted 2017-04-20 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections; acetyl-glycyl-asparagyl-glutaminyl-glutamyl-glutaminyl-valyl-seryl-prolyl-leucyl-threonyl-leucyl-leucyl-lysyl-lysyl-tryptophyl-cysteinyl-Alexa Fluoro 680 C2C2-maleimide conjugate; Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: A total of 13 participants will be recruited for this study. Prior to the first study research MRI scan, 3 volunteer participants will be scanned with a known breast malignancy (Group 1). These participants will not have hyperpolarized 13C pyruvate administered. They will be scanned with a 13C phantom in order to test the functionality of the 13C coil.
  Subsequently, up to 10 volunteer participants with breast cancer requiring NAC, between 18 and 80 years of age with pathology- and imaging-confirmed breast cancer requiring NAC will be studied (Group 2). Imaging confirmation involves highly suspicious masses on mammography and/or ultrasound. Pathology confirmation involves image-guided core biopsy of the suspicious mass.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hyperpolarized Pyruvate (13C) Injection (Active Comparator): The Participants in the active comparator arm will be injected with study drug Hyperpolarized Pyruvate (13C) Injection at a dose of 0.43/ml/kg.
  After the injection research, MRI will be done and images evaluated.
  Interventions: Drug: Hyperpolarized Pyruvate (13C) Injection; Drug: NAC
- Coil Testing (Placebo Comparator): Participants will receive an MRI with a 1 cm diameter plastic ball that contains 13C-urea that acts as test object. It provides a signal that is used to ensure that the MRI system is functioning properly.
  Interventions: Other: Coil Testing; Drug: NAC

INTERVENTIONS:
Drug: Hyperpolarized Pyruvate (13C) Injection — The new imaging method being tested in this study is called Metabolic MRI, which provides pictures of the metabolism occurring within cancer cells. It also involves injection of a contrast medicine, Hyperpolarized Pyruvate (13C) Injection, into the arm vein. The Participants in the active comparator arm will be injected with study drug Hyperpolarized Pyruvate (13C) Injection at a dose of 0.43/ml/kg.
  Other Names: Imaging Agent
  Arms: Hyperpolarized Pyruvate (13C) Injection
Other: Coil Testing — Participants will receive an MRI with a 1 cm diameter plastic ball that contains 13C-urea that will act as a test object. The test object provides a signal that will be used to ensure that the MRI system is functioning properly for participants in Group 2 . The plastic ball does not come in contact with you and there are no known risks associated with it.
  Other Names: Sentinel tabletop breast imaging coil
  Arms: Coil Testing
Drug: NAC — Participants will be receiving NAC as part of their clinical treatment.
  Other Names: Neoadjuvant Chemotherapy

SUMMARY:
Breast cancer is the second most common form of cancer in women and the most frequent cause of death. Despite breast screening programs, a substantial number of women are diagnosed with cancers greater than 2 cm in size or locally advanced disease, which is best treated with neoadjuvant chemotherapy (NAC) prior to surgery. Approximately 10% of women diagnosed with breast cancer annually will have locally advanced breast cancer, defined as stage III disease, where the cancer has either spread to regional lymph nodes and/or other tissue in the area of the breast, but not to distant sites. NAC offers the advantages of downstaging the disease, potentially reducing the extent of surgery. Presently, gadolinium enhanced MRI is the standard test used to monitor disease response to chemotherapy, and demonstrates changes in tumour size and extent between pre-NAC and post-NAC. Unfortunately, changes in tumour size may occur late in treatment regimen, thus producing false-negative results on early magnetic resonance imaging (MRI). Therefore, newer imaging techniques beyond anatomical imaging are needed to identify tumours that are unresponsive to chemotherapy and potentially change treatment plan early on to avoid significant morbidity associated with prolonged chemotherapy.

A novel MRI technique utilizing hyperpolarized pyruvate has the potential to detect pathophysiological response early in the treatment regimen and would therefore allow for earlier identification of nonresponders and subsequent early modification of treatment regimens, if necessary.

DETAILED DESCRIPTION:
Objectives:

Primary Objective To assess feasibility of of acquiring time resolved, 3D 13C pyruvate MR images of breast cancer requiring neoadjuvant chemotherapy after administration of hyperpolarized 13C pyruvate.

Secondary Objectives

1. To determine the diagnostic accuracy of time resolved, 3D 13C pyruvate MR imaging after administration of hyperpolarized 13C pyruvate for differentiating breast cancer from normal breast parenchyma.
2. To spatially correlate lactate seen on hyperpolarized 13C MR to anatomic imaging with conventional MRI.
3. To assess if hyperpolarized 13C pyruvate MR can differentiate between tumour necrosis versus viable tumour
4. To acquire statistical information to help design, fund, and power future clinical studies with larger patient populations.

Overall Study Design This is a pilot prospective, single-institution study in participants who will receive NAC. Participants will be first informed of the study by personnelle within the patient's circle of care. If the patient expresses interest in participating in the study, the study's Clinical Research Coordinator will approach the patient to provide further information, answer any questions, provide study documentation, as well as to obtain informed consent if agreeable. Clinical procedures will be completed at Sunnybrook Health Sciences Centre (SHSC) under the supervision of medically trained personnelle.

- Population: A total of 13 participants will be recruited for this study. Prior to the first study research MRI scan, we will scan up to 3 volunteer participants with a known breast malignancy (Group 1). These participants will not have hyperpolarized 13C pyruvate administered. They will be scanned with a 13C phantom in order to test the functionality of the 13C coil.

Subsequently, up to 10 volunteer participants with breast cancer requiring NAC, between 18 and 80 years of age with pathology- and imaging-confirmed breast cancer requiring NAC will be studied (Group 2). Imaging confirmation involves highly suspicious masses on mammography and/or ultrasound. Pathology confirmation involves image-guided core biopsy of the suspicious mass.

* Design: Each participant will receive one research MRI scan on the 3T MRI scanner prior to NAC. This visit will occur separately from the patient's clinical dynamic contrast enhanced (DCE) MRI.
* Scan Timing: The research MRI exam will be scheduled before the initiation of NAC, and within 5 days prior to, or following, the clinical MRI scan.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants of all ethnic groups/ race categories (age: between 18 and 80 years old)
* Radiographic diagnosis and pathologic confirmation of breast cancer
* Undergoing NAC prior to breast-conservation surgery (not applicable to the 3 participants not receiving the injection)
* Estimated survival more than 1 month
* Informed consent
* The participant will also be asked to complete the standard MRI safety screening questionnaire, prior to their research scan and participation in the study.
* Negative pregnancy test for females of child bearing potential
* Aspartate aminotransferase (AST) <31 U/L
* Alanine aminotransferase (ALT) <31 U/L
* Creatinine 44 - 106 umol/L

Exclusion Criteria:

* Contraindication to MRI or intravenous contrast agents
* Women that are pregnant or breastfeeding
* Participants weighing >136 kgs (weight limit for the scanner tables)
* Participants with pacemakers, cerebral aneurysm clips, shrapnel injury or implantable electronic devices not compatible with MRI.
* Pregnant
* Claustrophobia
* Inability to lie still for 45-60 minutes
* Participants with a high risk factor for nephrogenic systemic fibrosis (NFS), including renal failure on dialysis, heart disease, diabetes, single kidney, hypertension/hypotension, multiple myeloma, peripheral vascular disease, or taking of specific medications (loop diuretics, NSAIDs (within 7 days of research MRI), aminoglycosides, vancomycin, amphotericin B, chemotherapy, or immunosuppressants).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Time resolved, 3D 13C pyruvate MR images using MRI | 6 Months
  Feasibility of of acquiring time resolved, 3D 13C pyruvate MR images of breast cancer requiring neoadjuvant chemotherapy after administration of hyperpolarized 13C pyruvate.

SECONDARY OUTCOMES:
Accuracy of time resolved, 3D 13C pyruvate MR imaging using visual analysis of MRI images | 6 Months
  Diagnostic accuracy of time resolved, 3D 13C pyruvate MR imaging after administration of hyperpolarized 13C pyruvate for differentiating breast cancer from normal breast parenchyma.
Lactate Correlation using visual analysis of MRI Images | 6 Months
  Correlate lactate seen on hyperpolarized 13C MR to anatomic imaging with conventional MRI.
Visual differentiation between tumour necrosis versus viable tumour | 6 Months
  Differentiate between tumour necrosis versus viable tumour with Hyperpolarized 13C pyruvate MRI

CONTACTS AND LOCATIONS:
Overall Officials: Charles Cunningham, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No